CLINICAL TRIAL: NCT02081092
Title: Evaluation and Treatment Planning of Patients With PAP Using Thrive Ultra Short Echo Time MRI and CT
Acronym: PAP
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-7051
Record Dates: First submitted 2014-02-12; First posted 2014-03-07 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Alveolar Proteinosis
Keywords: PAP; Pulmonary Alveolar Proteinosis; Pulmonary; Patients
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary Alveolar Proteinosis (PAP): Patients diagnosis with Pulmonary Alveolar Proteinosis.

SUMMARY:
The purpose of this study is twofold: to assess routine cat scan (CT) imaging as a biomarker for removal of lipoprotein surfactant via lung lavage (where CT is the gold-standard imaging technique for density quantification), and to utilize a novel UTE MRI protocol to similarly quantify surfactant removal. This study will also serve to generate baseline scanning that may aid in developing analytical tools to evaluate and treat specific lung regions of patients with PAP.

DETAILED DESCRIPTION:
This study will evaluate x-ray CT as a biomarker for surfactant lavage removal and evaluate an UTE-Thrive MRI protocol at CCHMC as an imaging alternative to CT. Potential subjects who meet study criteria will be identified by the Pulmonary physicians at Cincinnati Children's Hospital Medical Center (CCHMC) and University of Cincinnati (UC) through their clinic patients. The study will include two research MRIs (one pre lavage and the second 24 to 72 hours after the first lung lavage) and if there is a clinical CT performed pre lavage, then one research CT will also be performed with the second research MRI. All image analysis will be quantitative. Whole-lung and regional density will be calculated and evaluated before and after lung lavage, for a quantification of changes in density in the left lung and right lung separately. Since the one lung will serve as control, it will allow precise error estimation (which we expect to be quite small and largely related to differences in lung volume). One purpose of this protocol is to further refine and develop ultra-short echo time (UTE) MRI techniques since Pulmonary Alveolar Proteinosis (PAP) patients may have multiple lavage sessions per year. A subject may be eligible to re-enroll to participate multiple times if the total number of research CTs for all enrollments is one or less for that subject.

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed PAP scheduled for lung lavage with double lumen endoscopy.

* Children patients ≥ 8 years of age
* Adult patients ≤ 75 years of age
* Medically stable as per the opinion of Bruce Trapnell, MD or Robert Wood, MD
* Patient and or parent consent obtained

Exclusion Criteria:

* Standard MRI exclusion criteria as set forth by the CCHMC Division of Radiology
* Pregnancy

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pulmonary Alveolar Proteinosis
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Comparing MRI's images pre and post whole lung lavage | 24 hours before lung lavage and 24-48 hours after lung lavage

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States